CLINICAL TRIAL: NCT02943109
Title: High Tech and High Touch (HT2): Transforming Patient Engagement Through Portal Technology at the Bedside
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ann McAlearney, Professor of Family Medicine and Executive Director, CATALYST, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HS024091 (AHRQ)
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Physician-Patient Relations; Inpatient Facility Diagnoses; Electronic Health Records; Outpatient
Keywords: patient portal; Health Information Technology; Electronic Health Records; Inpatient Care; Outpatient Care; Patient Engagement
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High tech, high touch (Experimental): Patient receives the full version of MyChart Bedside. Patient receives training/intervention from technology navigator
  Interventions: Other: High Touch; Other: High Tech
- Low tech, high touch (Experimental): Patient receives the non-interactional version of MyChart Bedside. Patient receives training/intervention from technology navigator
  Interventions: Other: High Touch; Other: Low Tech
- High tech, low touch (Experimental): Patient receives the full version of MyChart Bedside. Patient receives online training, only
  Interventions: Other: Low Touch; Other: High Tech
- Low tech, low touch (Experimental): Patient receives the non-interactional version of MyChart Bedside. Patient receives online training, only
  Interventions: Other: Low Touch; Other: Low Tech

INTERVENTIONS:
Other: High Touch — Participants receives an in person visit from an "technology navigator" who helps to explain the technology to the patient.
  Arms: High tech, high touch; Low tech, high touch
Other: Low Touch — Participants receives a visit from a "patient navigator" who helps to explain how to navigate the hospital system (active control).
  Arms: High tech, low touch; Low tech, low touch
Other: High Tech — Patient receives full-suite access to an inpatient patient portal with bi-directional communication enabled.
  Arms: High tech, high touch; High tech, low touch
Other: Low Tech — Patient receives a limited access version of the inpatient patient portal with bi-directional communication disabled.
  Arms: Low tech, high touch; Low tech, low touch

SUMMARY:
A large-scale randomized control trial (RCT) of the impact and use of an inpatient tablet-based patient portal embedded in a larger mixed methods study to examine changes in patient experiences and outcomes, and subsequent ambulatory patient portal usage.

DETAILED DESCRIPTION:
The appropriate use of technology to actively engage with patients who suffer from multiple chronic conditions, called multimorbidity, is one of the frontiers of both research and practice. For multimorbid patients, engagement in disease management activities is particularly critical, and evidence shows that enhanced patient self-management can lead to better control of chronic illness. One tool finding increasing use is the patient portal, and its pervasiveness is supported by virtue of its role as a component of the Meaningful Use criteria. A patient portal is a tethered personal health record (tPHR) that links to the patient's electronic health record, facilitating communication and engagement activities with healthcare providers. While most tPHRs have been focused on outpatient activities, a new class of tools focused on the inpatient experience has begun deployment in 2014.

In response, this study supports the conduct of the first, large-scale randomized control trial (RCT) of the impact and use of an inpatient tablet-based patient portal embedded in a larger mixed methods study to examine changes in patient experiences and outcomes, and subsequent ambulatory patient portal usage. The investigators aim to study how access to a patient portal tailored to the inpatient stay can improve patient experience and increase patient engagement by improving patients' perception of the process of care while in the hospital (patient experience), increasing patients' self-efficacy for managing their chronic conditions (patient engagement), and facilitating use of a patient portal for care management activities after discharge (patient engagement).

The study site is a world-class healthcare facility with the ability to provide access to a patient portal designed specifically for the inpatient experience, bridging to outside the hospital after discharge.

Currently, this inpatient technology exists in only one other hospital in the US, but the investigators expect that as inpatient PHRs become more readily available, the need for clarity on this issue will only increase. The investigator's evaluation is a mixed-methods design consisting of primary data collection through surveys and interviews throughout the study period, and secondary data collection from the electronic health record and health system metadata. This study will offer insight into a potentially important mechanism to facilitate patient self-management.

ELIGIBILITY:
Inclusion criteria:

* patient accepted MyChart Bedside tablet
* patient available in their room
* capable of providing informed consent

Exclusion criteria:

* Patient in a pilot unit where Full Tech was available prior to study start
* Patient was less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3782 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann S McAlearney, ScD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data types: Deidentified participant data.
  How to access data: Data may be requested from the PI via a request to ht2study@osumc.edu.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting date: 2023-07-01
  End date: 2027-06-30
Access Criteria: Who can access the data: Open to all requesters who provide a methodologically sound proposal whose use has also been approved by an independent review committee.
  Types of analyses: There are no a priori limits. Limits are based on approved proposals.
  Mechanisms of data availability: Secure Data transfer. Interested parties will be required to complete an institutional Data Use Agreement.

REFERENCES:
- [Background] McAlearney AS, Sieck CJ, Hefner JL, Aldrich AM, Walker DM, Rizer MK, Moffatt-Bruce SD, Huerta TR. High Touch and High Tech (HT2) Proposal: Transforming Patient Engagement Throughout the Continuum of Care by Engaging Patients with Portal Technology at the Bedside. JMIR Res Protoc. 2016 Nov 29;5(4):e221. doi: 10.2196/resprot.6355. PMID 27899338
- [Derived] Walker DM, Hefner JL, MacEwan SR, Di Tosto G, Sova LN, Gaughan AA, Huerta TR, McAlearney AS. Differences by Race in Outcomes of an In-Person Training Intervention on Use of an Inpatient Portal: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245091. doi: 10.1001/jamanetworkopen.2024.5091. PMID 38573634
- [Derived] McAlearney AS, Walker DM, Sieck CJ, Fareed N, MacEwan SR, Hefner JL, Di Tosto G, Gaughan A, Sova LN, Rush LJ, Moffatt-Bruce S, Rizer MK, Huerta TR. Effect of In-Person vs Video Training and Access to All Functions vs a Limited Subset of Functions on Portal Use Among Inpatients: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231321. doi: 10.1001/jamanetworkopen.2022.31321. PMID 36098967

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 3,782 enrolled participants, 2,892 met the study inclusion criteria and were randomized to one of the four study arms. Of those excluded:
  * 734 had an enrollment admission < 3 days;
  * 17 had no inpatient portal use on record;
  * 139 switched Tech assignment.
Period: Overall Study
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Started | 1242 | 470 | 905 | 275
Completed | 1242 | 470 | 905 | 275
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch | Total
Number analyzed (Participants) | 1242 | 470 | 905 | 275 | 2892
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [34 to 58] | 48 [36 to 60] | 47 [34 to 59] | 48 [36 to 60] | 47 [35 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 709 | 256 | 521 | 155 | 1641
  Male | 533 | 214 | 384 | 120 | 1251
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 976 | 368 | 675 | 202 | 2221
  Black | 225 | 81 | 186 | 58 | 550
  Other | 41 | 21 | 44 | 15 | 121
Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: units on a scale] — The Charlson Comorbidity Index is an assessment tool designed to predict long-term mortality. It is based on the concurrent presence of 17 morbidities, weighted for severity, and the age of the patient. Scores range between 0 and 37. Lower scores are better. A score of zero means no comorbidities were found.
  units on a scale | 1 [0 to 3] | 1 [0 to 3] | 2 [0 to 3] | 2 [0 to 3] | 1 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Inpatient Portal Use Frequency
Description: The count of MyChart Bedside (inpatient portal) sessions for the admission associated with study enrollment.
Time Frame: At hospital discharge.
Measure: Mean (Standard Deviation); unit: Inpatient portal sessions
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 1242 | 470 | 905 | 275
Inpatient portal sessions | 29 (31) | 21 (18) | 29 (36) | 20 (26)

2. Primary Outcome: Inpatient Portal Comprehensiveness of Use
Description: Based on the use of all available MyChart Bedside (inpatient portal) functions, a comprehensive inpatient portal user was one who used all three functions - for patients in the low tech assignment - or used eight or more functions - for patients in the high tech assignment.
Time Frame: At hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 1242 | 470 | 905 | 275
Participants | 697 | 292 | 253 | 104

3. Primary Outcome: Inpatient Portal Functions Proportion of Use
Description: For each MyChart Bedside (inpatient portal) function available to patients assigned to high tech, a proportion of total use is calculated for each patient as the sum of actions in a given function divided for the total sum of user actions during the hospital admission associated with study enrollment.
Time Frame: At hospital discharge.
Measure: Mean (Standard Deviation); unit: Proportion of total use
Arm/Group | High Tech, High Touch | High Tech, Low Touch
Number analyzed (Participants) | 1242 | 905
Proportion of total use
  Dining on Demand | 0.20 (0.17) | 0.22 (0.20)
  Tutorial | 0.16 (0.18) | 0.19 (0.22)
  To Learn | 0.02 (0.04) | 0.01 (0.05)
  My Health | 0.11 (0.15) | 0.10 (0.17)
  Happening Soon | 0.39 (0.23) | 0.37 (0.25)
  Notes | 0.00 (0.00) | 0.00 (0.00)
  Messages | 0.03 (0.04) | 0.03 (0.05)
  I Would Like | 0.00 (0.01) | 0.00 (0.01)
  MyChart | 0.03 (0.04) | 0.03 (0.04)
  Taking Care of Me | 0.05 (0.04) | 0.04 (0.05)

4. Primary Outcome: Patient Satisfaction With Care - Responses From Healthcare Professionals
Description: Questions from the satisfaction and experience domains of the 15-day Post-discharge surveys were used to assess patient satisfaction with their care. Answers to the following 5-point Likert scale survey item were explored: "In your most recent hospital experience, how satisfied were you with how well your healthcare professionals responded to your concerns? ". Responses were dichotomized to one "most positive" response versus all other responses.
Time Frame: 15 days after discharge
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Participants with positive response
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 197 | 76 | 93 | 30
Participants with positive response | 142 | 49 | 59 | 23

5. Primary Outcome: Patient Satisfaction With Care - Interactions With Healthcare Professionals
Description: Questions from the satisfaction and experience domains of the 15-day Post-discharge surveys were used to assess patient satisfaction with their care. Answers to the following 5-point Likert scale survey item were explored: "In your most recent hospital experience, how satisfied were you with the interactions you had with your healthcare professionals? ". Responses were dichotomized to one "most positive" response versus all other responses.
Time Frame: 15 days after discharge
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Participants with positive response
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 198 | 75 | 94 | 30
Participants with positive response | 150 | 50 | 59 | 22

6. Primary Outcome: Patient Satisfaction With Care - Responses From Healthcare Professionals
Description: Questions from the satisfaction and experience domains of the 6-month Post-discharge surveys were used to assess patient satisfaction with their care. Answers to the following 5-point Likert scale survey item were explored: "In the past 6 months, how satisfied were you with how well your healthcare professionals responded to your concerns? ". Responses were dichotomized to one "most positive" response versus all other responses.
Time Frame: 6 months after discharge
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Participants with positive response
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 222 | 105 | 185 | 46
Participants with positive response | 139 | 59 | 117 | 24

7. Primary Outcome: Patient Satisfaction With Care - Interactions With Healthcare Professionals
Description: Questions from the satisfaction and experience domains of the 6-month Post-discharge surveys were used to assess patient satisfaction with their care. Answers to the following 5-point Likert scale survey item were explored: "In your most recent hospital experience, how satisfied were you with the interactions you had with your healthcare professionals? ". Responses were dichotomized to one "most positive" response versus all other responses.
Time Frame: 6 months after discharge
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Participants with positive response
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 227 | 106 | 189 | 47
Participants with positive response | 153 | 63 | 127 | 33

8. Primary Outcome: Patient Involvement With Care - Questions About Health Management
Description: Questions from the involvement with care domain of the 15-day Post-discharge surveys were used to assess patient involvement with their care. Answers to the following 5-point Likert scale survey item were explored: "All of my questions about managing my health, including my medications, were addressed before I left the hospital.". Responses were dichotomized to one "most positive" response versus all other responses.
Time Frame: 15 days after discharge.
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Participants with positive response
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 153 | 58 | 184 | 58
Participants with positive response | 112 | 37 | 118 | 37

9. Primary Outcome: Patient Involvement With Care - Finding Answers to Health Management Questions
Description: Questions from the involvement with care domain of the 15-day Post-discharge surveys were used to assess patient involvement with their care. Answers to the following multiple-choice survey item were explored: "If you had a question about your care while you were in the hospital, what steps did you take to find an answer? (mark all that apply)".
Time Frame: 15 days after discharge.
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Patients
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 233 | 86 | 106 | 32
Patients
  I asked my doctor | 167 | 66 | 82 | 26
  I asked a nurse | 217 | 76 | 94 | 29
  I asked hospital staff | 58 | 26 | 30 | 10
  I searched online | 70 | 21 | 39 | 9
  Other | 16 | 5 | 7 | 1
  I did not have questions | 8 | 1 | 3 | 1

10. Primary Outcome: Patient Involvement With Care - Tablet's Activities
Description: Questions from the involvement with care domain of the 15-day Post-discharge surveys were used to assess patient involvement with their care. Answers to the following multiple-choice survey item were explored: "What kind of activities did you use the table for? (mark all that apply)".
Time Frame: 15 days after discharge.
Population: Patients who responded to the selected survey item.
Measure: Number; unit: Patients
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 233 | 85 | 104 | 32
Patients
  Email | 33 | 9 | 14 | 5
  Research health issues | 114 | 34 | 52 | 15
  Social media | 41 | 9 | 22 | 9
  Watch movies/TV | 20 | 6 | 7 | 3
  Communicate with family | 20 | 5 | 9 | 3
  Play games | 65 | 27 | 31 | 14
  MyChart Bedside | 217 | 73 | 93 | 26
  None of the above | 8 | 6 | 5 | 3

11. Secondary Outcome: Outpatient Portal Adoption
Description: MyChart (outpatient portal) accounts activated by participants after their enrollment in the study (based on log file analysis).
Time Frame: 3 months post-discharge
Population: Participants without an active outpatient portal account at the time of their enrollment in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 688 | 290 | 508 | 179
Participants | 218 | 66 | 126 | 29

12. Secondary Outcome: Outpatient Portal Frequency of Use
Description: Count of MyChart (outpatient portal) sessions (based on log file analysis).
Time Frame: 3 months post-discharge
Population: Patients with an active outpatient portal account; either predating their participation in the study (Previous users) or activated after study enrollment (New users).
Measure: Mean (Standard Error); unit: Outpatient portal sessions
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 772 | 246 | 523 | 125
Outpatient portal sessions
  New users: number analyzed (Participants) | 218 | 66 | 126 | 29
  New users | 21 (32) | 19 (21) | 17 (25) | 20 (29)
  Previous users: number analyzed (Participants) | 554 | 180 | 397 | 96
  Previous users | 35 (41) | 41 (44) | 38 (48) | 37 (38)

13. Secondary Outcome: Self-Efficacy
Description: 5-point Likert scale built on the participant responses to 6 self-efficacy-related items from the admission survey. Self-efficacy measures the belief in one's capacity to complete a task, rather than the relevant skills possessed. Scale developed on the basis of Bandura, A. (2006). Guide for constructing self-efficacy scales. In F. Pajares & T. Urdan (Eds.). Self-Efficacy Beliefs of Adolescent. Greenwich, CT: Information Age Publishing, pp. 307-337.
  Self-Efficacy scale:
  * min value: 1;
  * max value: 5;
  * higher scores are better outcomes.
Time Frame: Baseline
Population: Patients who completed the self-efficacy section of the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 864 | 349 | 626 | 184
score on a scale | 4.3 (0.6) | 4.3 (0.5) | 4.3 (0.6) | 4.2 (0.6)

14. Secondary Outcome: Self-Efficacy
Description: as for outcome 13
Time Frame: 15 days post-discharge
Population: Patients who completed the self-efficacy section of the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 228 | 86 | 102 | 32
score on a scale | 4.5 (0.5) | 4.5 (0.5) | 4.4 (0.7) | 4.4 (0.7)

15. Secondary Outcome: Self-Efficacy
Description: as for outcome 13
Time Frame: 6 months post-discharge
Population: Patients who completed the self-efficacy section of the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
Number analyzed (Participants) | 269 | 118 | 214 | 55
score on a scale | 4.3 (0.6) | 4.3 (0.5) | 4.3 (0.6) | 4.2 (0.7)

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | High Tech, High Touch | Low Tech, High Touch | High Tech, Low Touch | Low Tech, Low Touch
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT02943109/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT02943109/SAP_001.pdf
  • Informed Consent Form (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02943109/ICF_002.pdf